CLINICAL TRIAL: NCT02394509
Title: HOBSCOTCH Phase II: A Pragmatic Study of HOBSCOTCH in New England.
Brief Title: HOBSCOTCH Phase II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Barbara Jobst, Staff Physician, Neurology, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: D12217 Phase II
Record Dates: First submitted 2015-03-06; First posted 2015-03-20 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Epilepsy
Keywords: Epilepsy Memory Problems; Self-Management
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- HOBSCOTCH-IP (in person) (Experimental): Participants will receive the HOBSCOTCH intervention consisting of a first session conducted in-person, 3 weekly followed by 3 bi-weekly telephone coaching sessions, and a final session conducted in-person.
  Interventions: Behavioral: Home Based Self-management and Cognitive Training Changes lives (HOBSCOTCH)
- HOBSCOTCH-V (virtual) (Experimental): Participants will receive the HOBSCOTCH intervention consisting of a first session conducted virtually, 3 weekly followed by 3 bi-weekly telephone coaching sessions, and a final session conducted virtually.
  Interventions: Behavioral: Home Based Self-management and Cognitive Training Changes lives (HOBSCOTCH)
- Control (Other): Participants will be wait listed and given an option whether they prefer to enroll into HOBSCOTCH-IP or HOBSCOTCH-V. Subjects in Group 3 will receive HOBSCOTCH following a 6 month wait period.
  Interventions: Behavioral: Home Based Self-management and Cognitive Training Changes lives (HOBSCOTCH)

INTERVENTIONS:
Behavioral: Home Based Self-management and Cognitive Training Changes lives (HOBSCOTCH) — HOBSCOTCH is a home-based self-management program to treat cognitive symptoms and improve quality of life, while minimizing the barriers of access to care. The program is based on Problem Solving Therapy (PST) and teaches problem solving strategies and compensatory mechanisms to help manage cognitive dysfunction and enhance quality of life.

SUMMARY:
The purpose of this study is to determine the feasibility and efficacy of the home-based cognitive self-management program "HOBSCOTCH" delivered at four New England medical centers. It will test the long-term impact and cost-effectiveness of HOBSCOTCH, and whether it can be delivered from a distance utilizing e-health tools for parts of the program.

DETAILED DESCRIPTION:
HOBSCOTCH (Home Based Self-management and Cognitive Training Changes lives) is a home-based self-management program to treat cognitive symptoms and improve quality of life, while minimizing the barriers of access to care. The program is based on Problem Solving Therapy (PST) and teaches problem solving strategies and compensatory mechanisms to help manage cognitive dysfunction and enhance quality of life.

HOBSCOTCH Phase II is a replication study of the original HOBSCOTCH study, designed to translate the findings of HOBSCOTCH into a real world setting. This is a multi-center study, with the HOBSCOTCH intervention being implemented at four epilepsy clinics in New England.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* Confirmed diagnosis of epilepsy, with controlled or uncontrolled seizures
* Subjective memory complaints
* No changes in antiepileptic and antidepressant medication regimen for 1 month, however brief discontinuation of antiepileptic medicine for inpatient video EEG evaluation is acceptable
* Literate
* Telephone access

Exclusion Criteria:

* Subjects age 66-70 with a mention of a dementing illness in their medical record
* Severe mental disability or estimated IQ less than 70
* Significant visual impairment precluding reading or writing
* No reliable telephone access

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life | Baseline and months: 3, 6, 9, 12, 15
  We will be using Quality of Life in Epilepsy (QOLIE-31). This validated tool contains 16 multi-item scales which assess health related quality of life, emotional well-being, memory and attention deficits, medication effects, seizure control, psychosocial functioning, and health perception
Change in Healthcare Utilization | Baseline and months: 3, 6, 9, 12, 15
  We will be using the Healthcare Utilization in Epilepsy (HCU-E). This validated survey is concordant with billing data. It assesses seizure frequency and whether the subject had received any of the following services because of their epilepsy over the past 3 months: hospital ER services, general practice or family doctor visits, neurologist or epilepsy specialist visits, and overnight hospital inpatient stay.

SECONDARY OUTCOMES:
Change in Depression | Baseline and months: 3, 6, 9, 12, 15
  We will be using the Patient Health Questionnaire (PHQ-9). The PHQ-9 is a brief 9-item validated depression scale.
Change in Cognition | Baseline and months: 3, 6, 9, 12, 15
  We will be using a modified version of the Brief Test of Adult Cognition by Telephone (BTACT). This is a modified version of a validated psychometric instrument that can be delivered over the phone in 20 minutes. It includes measures of episodic memory, working memory, reasoning, verbal fluency and executive function.
Change in Self-Management Practices | Baseline and months: 3, 6, 9, 12, 15
  We will be using the Epilepsy Self-Management Scale (ESMS). This is a 38 item scale that assesses use of epilepsy self-management practices.
Change in Cognitive Function | Baseline and months: 3, 6, 9, 12, 15
  We will be using the Cognitive Function sub-scale of the NeuroQOL. This is a brief validated tool developed by the NIH for use in patients with neurological disease.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara C Jobst, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center and Dartmouth College
Locations (4):
- United States (4):
  - Maine Medical Center, Portland, Maine
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Dartmouth-Hitchcock Medical Center in Lebanon, NH, Lebanon, New Hampshire
  - University of Vermont Medical Center, Burlington, Vermont

REFERENCES:
- [Derived] Streltzov NA, Schmidt SS, Schommer LM, Zhao W, Tosteson TD, Mazanec MT, Kiriakopoulos ET, Chu F, Henninger HL, Nagle K, Roth RM, Jobst B. Effectiveness of a Self-Management Program to Improve Cognition and Quality of Life in Epilepsy: A Pragmatic, Randomized, Multicenter Trial. Neurology. 2022 May 24;98(21):e2174-e2184. doi: 10.1212/WNL.0000000000200346. Epub 2022 Apr 6. PMID 35387855